CLINICAL TRIAL: NCT05820932
Title: Plasma Amyloid-beta 42/40 to Predict Cognitive Decline From Androgen Deprivation Therapy in Prostate Cancer: a Prospective Observational Study
Brief Title: Predicting Cognitive Decline From Androgen Deprivation Therapy
Acronym: ABC
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 22806; NCI-2023-02192 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: Cognitive decline; Cognitive functioning
MeSH Terms: conditions — Prostatic Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants with prostate cancer, ADT (ADT Cohort): This group is comprised of adult men with hormone-sensitive prostate cancer who are starting androgen deprivation therapy as part of standard of care prostate cancer (not as part of this protocol).
  Interventions: Genetic: Blood-based assay; Diagnostic Test: Cognitive assessments; Other: Quality of Life Surveys
- Participants in remission, No ADT (Prostate cancer Control (PC) Cohort)): This group is comprised of adult men who are in remission from prostate cancer who have never received ADT.
  Interventions: Genetic: Blood-based assay; Diagnostic Test: Cognitive assessments; Other: Quality of Life Surveys
- Partners of Participants: Study partner participants will also be recruited
  Interventions: Other: Quality of Life Surveys

INTERVENTIONS:
Genetic: Blood-based assay — Blood samples will be collected
  Groups: Participants in remission, No ADT (Prostate cancer Control (PC) Cohort)); Participants with prostate cancer, ADT (ADT Cohort)
Diagnostic Test: Cognitive assessments — Cognitive assessments will be both participant- and partner-reported
  Groups: Participants in remission, No ADT (Prostate cancer Control (PC) Cohort)); Participants with prostate cancer, ADT (ADT Cohort)
Other: Quality of Life Surveys — Participant-reported Quality of Life Surveys
  Other Names: QoL Surveys

SUMMARY:
Androgen Deprivation Therapy (ADT) is associated with cognitive impairment and dementia in men with prostate cancer. Pre-clinical data suggest that ADT-induced hypogonadism leads to accumulation of beta-amyloid plaques in the hippocampus, a pathological hallmark of Alzheimer's Disease (AD). Neuroimaging Functional magnetic resonance imaging (fMRI) studies also demonstrate that ADT decreases metabolic activity in the parietal, occipital, and prefrontal cortices. Multiple prospective cohort and population-based clinical studies have been conducted to test the association between ADT and cognitive impairment and/or dementia.

Plasma biomarkers have been developed to predict brain amyloidosis, a key pathological feature of AD and a risk factor for developing dementia due to AD. The advantage of a blood-based assay is the lower cost, invasiveness, and time compared to cerebrospinal fluid (CSF) and Positron Emission Tomography (PET)-based biomarkers.

DETAILED DESCRIPTION:
This is a single-site, non-randomized prospective observational study of men with prostate cancer.

PRIMARY OBJECTIVE:

I. To evaluate whether baseline plasma Amyloid-beta 42/40 (Aβ42/40) ratio is associated with cognitive decline in men upon starting ADT.

SECONDARY OBJECTIVE:

I. To evaluate whether ADT is associated with a decline in plasma Aβ42/40 ratio.

II. To evaluate whether intensified ADT (iADT) receipt is associated with greater cognitive decline compared to ADT.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants-

* Age 18 years or greater.
* Fluent in reading, listening to, and writing English.
* Current or prior diagnosis of prostate adenocarcinoma based on a pathology report or as documented in a medical oncology, urology, or radiation oncology note.
* Access and ability to use a computer or mobile device with Internet connectivity to complete study procedures.
* Telephone Montreal Cognitive Assessment (T-MoCA) of 16 or greater.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (documented within past 3 months, otherwise patient-reported).

Study partner participants-

* Age 18 years or greater
* Fluent in reading, listening to, and writing English
* Identified by patient participant as a person who knows patient participant well, like a friend, family member or spouse.
* Access and ability to use a computer or mobile device with internet connectivity to complete study procedures.

Only the ADT cohort-

* Anticipated to start ADT, which includes one of the following two treatments

  * Gonadotropin-releasing hormone (GnRH) agonist (e.g., leuprolide, goserelin, and others).
  * GnRH antagonist (i.e., degarelix or relugolix).
* Anticipated to remain on ADT for at least 12 months.
* Concurrent first-generation anti-androgens (e.g., bicalutamide, flutamide, nilutamide) and novel androgen-signaling inhibitors (e.g., abiraterone, enzalutamide, and apalutamide) are allowed.
* Concurrent radiation is allowed.

Only the PC cohort-

* Has completed definitive local therapy (radical prostatectomy or radiation therapy) for localized prostate cancer at least 6 months prior to screening.
* For radical prostatectomy: undetectable prostate-specific antigen (PSA) within 12 months of screening.
* For radiation therapy: last PSA of < 2.0 within 12 months of screening.

Exclusion Criteria:

Patient Participants-

* Small cell prostate carcinoma (pure or mixed).
* Receipt of ADT (GnRH agonist, GnRH antagonist, 1st-generation anti-androgen, or novel androgen signaling inhibitor) within 6 months before screening. ADT >6 months prior to screening is allowed provided testosterone has recovered to 100 ng/ml or greater.
* Concurrent or anticipated (at any point during first 12 months of ADT) non-hormonal, antineoplastic systemic therapy, such as chemotherapy.
* Testosterone <100 ng/ml.
* Prior or concurrent brain metastases (no prior or screening imaging is required).
* Major neurocognitive or psychiatric disorders, such as dementia or schizophrenia.
* Prior or concurrent malignancy other than prostate cancer whose natural history or treatment has the potential to interfere with study assessments.

Study partner participants-

* None.

Only the ADT cohort-

* None.

Only the PC cohort-

* Any prior, concurrent, or anticipated use of any hormonal systemic therapy, including GnRH agonist, GnRH antagonist, 1st-generation anti-androgen, or novel androgen signaling inhibitor.
* Any known or prior history of M1 prostate cancer (no screening imaging required).
* Current or prior biochemical recurrence following American Urological Association guidelines for radical prostatectomy or American Society for Therapeutic Radiology and Oncology (ASTRO) guidelines for radiation therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with prostate cancer and partners of participants. The analysis population will consist of participants who complete baseline plasma Aβ42/40 and apolipoprotein E4 (APOE4) collection and the cognitive assessments at baseline and at least 3 months.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with cognitive decline (ADT cohort) | Up to 12 months
  Proportion with cognitive decline, defined as a decrease in >=1 neurocognitive test after ADT by >=1 standard deviation (SD) compared to baseline.
Mean cognitive decline (ADT cohort) | Up to 12 months
  The Z-scores of each cognitive test after receiving ADT will be calculated as a repeated measure.
Proportion of participants with cognitive impairment after ADT (ADT Cohort) | Up to 12 months
  Proportion of participants with cognitive impairment after receiving ADT, defined as a score of >=1 SD below normative mean score (i.e., PC control) in >=1 of the neurocognitive tests given during the course of ADT therapy.

SECONDARY OUTCOMES:
Change in mean plasma Aβ42/40 ratio | Up to 12 months
  Change in mean plasma Aβ42/40 ratio for the ADT cohort at 12 months will be compared to that of the PC control cohort
Mean cognition score | Up to 12 months
  The Z-scores of each cognitive test will be calculated as a repeated measure.
Mean study partner-reported cognition score | Up to 12 months
  The Z-scores of each cognitive test will be calculated as a repeated measure.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kwon, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No